CLINICAL TRIAL: NCT05426304
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Agomelatine in the Prevention of Poststroke Depression
Brief Title: Prophylactic Effects of Agomelatine for Poststroke Depression
Acronym: PRAISED
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jinsheng Zeng, MD, PhD, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRAISED
Record Dates: First submitted 2022-05-02; First posted 2022-06-21 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Depression; Acute Ischemic Stroke
Keywords: poststroke depression, prevention, agomelatine
MeSH Terms: conditions — Depression; Ischemic Stroke | interventions — agomelatine; Placebo Effect

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Agomelatine (Experimental): The Agomelatine group will be received agomelatine (25 mg/day) for 180 days.
  Interventions: Drug: Agomelatine
- Placebo (Placebo Comparator): The Placebo group will be received placebo (25 mg/day) for 180 days.
  Interventions: Drug: Placebo Tablets

INTERVENTIONS:
Drug: Agomelatine — agomelatine 25 mg/day for 180 days
  Other Names: Agomelatine Tablets
  Arms: Agomelatine
Drug: Placebo Tablets — placebo 25 mg/day for 180 days
  Other Names: Placebo Placebo
  Arms: Placebo

SUMMARY:
The incidence of depression in stroke patients with frontal lobe involvement was reported to be as high as 42%. Agomelatin, a type 1/2 melatonin receptor agonist and serotonin 2C receptor antagonist, is effective in treatment of depression, but whether it can prevent poststroke depression (PSD) remains unknown. The PRAISED trial is a multicenter, randomized, double-blind trial and is designed to evaluate the efficacy and safety of agomelatine in the prevention of PSD in stroke patients with frontal lobe involvement. The primary outcome is the rate of post-stroke depression for 180 days.

DETAILED DESCRIPTION:
This PRAISED trial is a multicenter, randomized, double-blind trial to evaluate the efficacy and safety of agomelatine in the prevention of PSD in patients with acute ischemic stroke. The sample size is 420. The participants will be randomized to receive a 6-month treatment of agomelatine 25mg/d or placebo 25mg/d. The primary end point is the proportion of PSD within 180 days. PSD is defined as the Hamilton Depression Rating Scale-17 (HAMD-17) ≥7 or diagnosis of depression by the Diagnostic and Statistical Manual of mental disorders-V (DSM-V). The second end point are rate of recurrence of ischemic stroke within 90 days, modified Rankin Scale (mRS), National Institutes of Health Stroke Scale (NIHSS), vascular death, transient ischemic attack (TIA)/stroke or myocardial infarction during the 6-months, cognitive function(Mini Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA)), Pittsburgh Sleep Quality Index (PSQI), Fatigue Severity Scale (FSS), Epworth Sleepiness Scale (ESS), Stroke Specific Quality Of Life (SS-QOL) scale, adherence to medication, adverse events. The study consists of five visits including the day of randomization, day 14±3 days, day 28±3 days, day 90±7 days, day 180±7 days.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18~75 years;
2. within 7 days after stroke onset;
3. CT or MRI showed lesions involving the frontal lobe;
4. mRS≤2 before onset for recurrent ischemic stroke;
5. HAMD-17<8 before enrollment;
6. NIHSS<16;
7. be consious and able to complete the relevant assessment scales.

Exclusion Criteria:

1. hemorrhagic stroke;
2. with major depressive disorder, or have taken antidepressants within 30 days before stroke onset, or HAMD-17 ≥8;
3. with other mental illnesses;
4. history of drug abuse or alcohol dependence in the past 1 year
5. with life-threatening illnesses or disorders which may affect the completion of the relevant assessment scale (e.g., hearing, language, visual impairment, etc.)
6. with cognitive impairment who cannot complete the relevant assessment scale
7. with serious neurodegeneration diseases (such as Parkinson's disease, Alzheimer's disease, etc.)
8. infection or carriers of hepatitis B virus (HBV) or hepatitis C virus (HCV)
9. serum ALT level ≥ 2 times of the upper limit of the reference interval or TBIL level > 1.5 times of the upper limit of the reference interval
10. renal dysfunction (creatinine clearance < 90 ml/min/1.73 m2)
11. allergic to or contra-indicated to agomelatine
12. lactose intolerance
13. pregnant or breast-feeding women
14. withdraw from other clinical trials within 4 weeks or participating in other clinical trials
15. unsuitable for inclusion considered by the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
rate of PSD within 180 days | 180 days
  PSD is defined as Hamilton Depression Rating Scale-17 (HAMD-17) ≥7 or diagnosis of depression by DSM-V.

SECONDARY OUTCOMES:
rate of recurrence of ischemic stroke within 90 days | 90±7 days
  1. Acute onset of focal neurological deficit, a few can be comprehensive neurological deficit. 2. Brain CT/MRI confirms the corresponding infarct focus in the brain, or the symptoms and signs continue for more than 24h, or cause death within 24h. 3. Exclude non-ischemic causes.
  2. brain ct/mri confirmed the corresponding infarct focus in the brain, or the symptoms and signs continued for more than 24h, or caused death within 24h.
  3. exclude non ischemic causes.
variation of HAMD-17 score from baseline | 14±3 days, 28±3 days, 90±7 days, and 180±7 days
  range from 0 to 50; the higher, the worse
rate of sleep disorder | 180 days
  range from 0 to 21; > 7, having sleep disorder
variation of Pittsburgh Sleep Quality Index (PSQI) score from baseline | 14±3 days, 28±3 days, 90±7 days and 180±7 days
  range from 0 to 21; the higher, the worse; > 7, having sleep disorder
variation of Stroke Specific Quality of Life (SS-QOL) score from baseline | 28±3 days, 90±7 days, and 180±7 days
  range from 50 to 248; the higher, the better
variation of Modified Rankin Scale (mRS) score from baseline | 28±3 days, 90±7 days and 180±7 days
  range from 0 to 5; the higher, the worse
variation of National Institutes of Health Stroke Scale (NIHSS) from baseline | 28±3 days, 90±7 days and 180±7 days
  range from 0 to 42; the higher, the worse
variation of Montreal Cognitive Assessment (MOCA) from baseline | 28±3 days, 90±7 days, and 180±7 days
  range from 0 to 30; the lower, the worse
variation of Mini Mental State Examination (MMSE) score from baseline | 28±3 days, 90±7 days, and 180±7 days
  range from 0 to 30; the lower, the worse
variation of Epworth Sleepiness Scale (ESS) from baseline | 28±3 days, 90±7 days, and 180±7 days
  range from 9 to 63; the higher, the worse
rate of all-caused mortality | 180 days
  death due to all causes
variation of Fatigue Severity Scale (FSS) from baseline | 28±3 days, 90±7 days, and 180±7 days
  range from 0 to 24; >=24, having drowsiness tendency
rate of vascular events | 180 days
  defined as the composite of stroke, transient ischemic attack (TIA), myocardial infarction and vascular death
rate of liver injury | 28±3 days, 90±7 days
  defend as the level of ALT 2 times higher than the upper limit of normal range

CONTACTS AND LOCATIONS:
Overall Officials: Jinsheng Zeng, Study Chair — First Affiliated Hospital, Sun Yat-Sen University

REFERENCES:
- [Background] Zhao FY, Yue YY, Li L, Lang SY, Wang MW, Du XD, Deng YL, Wu AQ, Yuan YG. Clinical practice guidelines for post-stroke depression in China. Braz J Psychiatry. 2018 Jul-Sep;40(3):325-334. doi: 10.1590/1516-4446-2017-2343. Epub 2018 Feb 1. PMID 29412338
- [Background] Hackett ML, Pickles K. Part I: frequency of depression after stroke: an updated systematic review and meta-analysis of observational studies. Int J Stroke. 2014 Dec;9(8):1017-25. doi: 10.1111/ijs.12357. Epub 2014 Aug 12. PMID 25117911
- [Background] Robinson RG, Jorge RE. Post-Stroke Depression: A Review. Am J Psychiatry. 2016 Mar 1;173(3):221-31. doi: 10.1176/appi.ajp.2015.15030363. Epub 2015 Dec 18. PMID 26684921
- [Background] Villa RF, Ferrari F, Moretti A. Post-stroke depression: Mechanisms and pharmacological treatment. Pharmacol Ther. 2018 Apr;184:131-144. doi: 10.1016/j.pharmthera.2017.11.005. Epub 2017 Nov 9. PMID 29128343
- [Background] Feng C, Fang M, Liu XY. The neurobiological pathogenesis of poststroke depression. ScientificWorldJournal. 2014 Mar 4;2014:521349. doi: 10.1155/2014/521349. eCollection 2014. PMID 24744682
- [Background] Gu J, Huang H, Chen K, Huang G, Huang Y, Xu H. Are they necessary? Preventive therapies for post-stroke depression: A meta-analysis of RCTs. Psychiatry Res. 2020 Feb;284:112670. doi: 10.1016/j.psychres.2019.112670. Epub 2019 Oct 31. PMID 31740211
- [Background] Kim JS, Lee EJ, Chang DI, Park JH, Ahn SH, Cha JK, Heo JH, Sohn SI, Lee BC, Kim DE, Kim HY, Kim S, Kwon DY, Kim J, Seo WK, Lee J, Park SW, Koh SH, Kim JY, Choi-Kwon S; EMOTION investigators. Efficacy of early administration of escitalopram on depressive and emotional symptoms and neurological dysfunction after stroke: a multicentre, double-blind, randomised, placebo-controlled study. Lancet Psychiatry. 2017 Jan;4(1):33-41. doi: 10.1016/S2215-0366(16)30417-5. PMID 28012485
- [Background] FOCUS Trial Collaboration. Effects of fluoxetine on functional outcomes after acute stroke (FOCUS): a pragmatic, double-blind, randomised, controlled trial. Lancet. 2019 Jan 19;393(10168):265-274. doi: 10.1016/S0140-6736(18)32823-X. Epub 2018 Dec 5. PMID 30528472
- [Background] Williams LS, Kroenke K, Bakas T, Plue LD, Brizendine E, Tu W, Hendrie H. Care management of poststroke depression: a randomized, controlled trial. Stroke. 2007 Mar;38(3):998-1003. doi: 10.1161/01.STR.0000257319.14023.61. Epub 2007 Feb 15. PMID 17303771
- [Background] Robinson RG, Jorge RE, Moser DJ, Acion L, Solodkin A, Small SL, Fonzetti P, Hegel M, Arndt S. Escitalopram and problem-solving therapy for prevention of poststroke depression: a randomized controlled trial. JAMA. 2008 May 28;299(20):2391-400. doi: 10.1001/jama.299.20.2391. PMID 18505948
- [Background] Almeida OP, Waterreus A, Hankey GJ. Preventing depression after stroke: Results from a randomized placebo-controlled trial. J Clin Psychiatry. 2006 Jul;67(7):1104-9. doi: 10.4088/jcp.v67n0713. PMID 16889454
- [Background] Chollet F, Tardy J, Albucher JF, Thalamas C, Berard E, Lamy C, Bejot Y, Deltour S, Jaillard A, Niclot P, Guillon B, Moulin T, Marque P, Pariente J, Arnaud C, Loubinoux I. Fluoxetine for motor recovery after acute ischaemic stroke (FLAME): a randomised placebo-controlled trial. Lancet Neurol. 2011 Feb;10(2):123-30. doi: 10.1016/S1474-4422(10)70314-8. Epub 2011 Jan 7. PMID 21216670
- [Background] Tsai CS, Wu CL, Chou SY, Tsang HY, Hung TH, Su JA. Prevention of poststroke depression with milnacipran in patients with acute ischemic stroke: a double-blind randomized placebo-controlled trial. Int Clin Psychopharmacol. 2011 Sep;26(5):263-7. doi: 10.1097/YIC.0b013e32834a5c64. PMID 21811172
- [Background] Niedermaier N, Bohrer E, Schulte K, Schlattmann P, Heuser I. Prevention and treatment of poststroke depression with mirtazapine in patients with acute stroke. J Clin Psychiatry. 2004 Dec;65(12):1619-23. doi: 10.4088/jcp.v65n1206. PMID 15641866
- [Background] Berg A, Palomaki H, Lehtihalmes M, Lonnqvist J, Kaste M. Poststroke depression: an 18-month follow-up. Stroke. 2003 Jan;34(1):138-43. doi: 10.1161/01.str.0000048149.84268.07. PMID 12511765
- [Background] Quera-Salva MA, Lemoine P, Guilleminault C. Impact of the novel antidepressant agomelatine on disturbed sleep-wake cycles in depressed patients. Hum Psychopharmacol. 2010 Apr;25(3):222-9. doi: 10.1002/hup.1112. PMID 20373473
- [Background] Chern CM, Liao JF, Wang YH, Shen YC. Melatonin ameliorates neural function by promoting endogenous neurogenesis through the MT2 melatonin receptor in ischemic-stroke mice. Free Radic Biol Med. 2012 May 1;52(9):1634-47. doi: 10.1016/j.freeradbiomed.2012.01.030. Epub 2012 Feb 10. PMID 22330064